CLINICAL TRIAL: NCT06424912
Title: Vivifi's Treatment, BPH Treatment Via Vasculature Anastomosis of the Internal Spermatic Vein and Ligation of the Deferential Vein
Brief Title: Vivifi's Treatment, BPH Treatment Via Vasculature Anastomosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vivifi Medical (Industry)
Collaborators: RQM+ (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP-001
Record Dates: First submitted 2024-05-13; First posted 2024-05-22 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Benign Prostatic Hyperplasia; Varicocele Grade II; Varicocele Grade III
Keywords: BPH; Varicocele
MeSH Terms: conditions — Prostatic Hyperplasia; Varicocele

STUDY DESIGN:
Intervention Model Description: Prospective, non-randomized first-in-man study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Group (Experimental): Subjects undergo Vivifi's surgical procedure for treatment of BPH.
  Interventions: Procedure: Vivifi's Surgical Procedure

INTERVENTIONS:
Procedure: Vivifi's Surgical Procedure — Subjects undergo Vivifi's surgical procedure for treatment of BPH. The study procedure will be performed in the operating room, under general anesthesia.
  Subject will undergo a bilateral anastomosis of the internal spermatic vein to the inferior epigastric vein and ligation of the deferential vein via bilateral inguinal/subinguinal incision.
  The investigators can use of a coupler with appropriate ring size (to be measured intra-operatively based on vessel size) to perform the vascular anastomosis and standard sutures for ligation. The coupler is an FDA approved commercial device. Alternatively, the anastomosis can also be performed using sutures. Incision closure will proceed per institution standard of care.

SUMMARY:
The study objective is to evaluate the safety and feasibility of the Vivifi's Treatment.

The Vivifi's Treatment presents an innovative approach for addressing benign prostatic hyperplasia (BPH) as well as clinical/subclinical varicoceles in men. The scientific rationale for conducting this study is to assess the safety and feasibility of the Vivifi's Treatment (a surgical procedure) as a therapeutic intervention for patients with BPH.

DETAILED DESCRIPTION:
Current BPH treatments fall into two major categories:

1. Surgical removal/destruction of prostatic tissues:

   1. Transurethral resection of the prostate (TURP)
   2. Holmium laser enucleation of the prostate (HoLEP)
   3. Aquablation - (Procept)
   4. Prostatic artery embolization (PAE)
2. Minimally-invasive Surgical Therapies (MISTs)

   1. Itind (now Olymus)
   2. Urolift (now Teleflex)
   3. Rezum (now Boston Scientific)
   4. TUNA
   5. Zenflow (in trials)
   6. Butterfly Medical (in trials)

The solutions in the first category rely in removing or destroying prostatic tissue. Though effective at reducing urinary symptoms, this damage to the tissue can cause a number of complications. The "non-surgical" solutions fall into the second category. One of the best-studied of these, Urolift, is an implant-based therapy, using internal sutures that are deployed though the urethra that pull the prostatic tissue away from the urethra lumen, repristinating urethral patency. A significant percentage of cases show recurrence of symptoms due to the fact that the prostate continues to grow. Looking at the currently available treatment options, the longer-lasting surgical procedure (group 1). Group 1 procedures, especially TURP, remain "the gold standard" by which all other BPH treatment options are measured.

The Vivifi's Treatment aims to fill the therapeutic gap between the two-category approaches by offering patients a less invasive surgical approach that (1) fixes the root cause of the problem, guaranteeing long lasting effects and (2) does not cause any damage to the prostatic tissue and urethra, thereby preventing the side effects mentioned above. By replumbing a faulty localized vasculature, the Vivifi's technology leverage years of safety data for anastomotic coupling rings enabling it for vascular surgical approaches. These initial clinical studies will prove that this totally novel treatment approach to BPH is safe.

ELIGIBILITY:
Inclusion Criteria:

1. Male 40-75 years of age
2. Diagnosed with Benign prostatic hyperplasia (BPH)
3. Prostate volume: ≥ 30 ≤ 120 cc measured by transrectal ultrasound
4. Signed the study informed consent form (ICF)
5. Presence of Lower Urinary Tract Symptoms (LUTS) measured by International Prostate Symptoms Score (IPSS) greater than 12
6. Presence of clinical varicocele (preferably grade II or III - Dubin & Amelar.

Exclusion Criteria:

1. Patients with prior history of spermatic vein or pampiniform plexus related surgeries or impairment, or vasectomy
2. Previous invasive prostate intervention (TURP, laser, ablation, prostate artery embolization, etc.)
3. Prostate with large intravesical median lobe
4. Patients with sub-clinical varicocele
5. Post-void residual volume (PVR) > 110ml
6. IPSS (International Prostate Symptoms Score) >24
7. Patients with clinical history of chronic prostatitis.
8. Patients with clinical history of urinary retention with previous need for catheterization (prior 30 days).
9. Major neurological conditions such as Alzheimer's, Parkinson, Multiple sclerosis, ALS, spinal cord injury
10. Patients that can not be under general anesthesia
11. Patients on blood thinners, or with coagulation related issues, TTP
12. Prior pelvic floor surgery or condition such as inguinal hernia, mesh, etc
13. History of cancer in genitourinary system, which is not considered being cured. A potential participant is considered cured if there has been no evidence of cancer within five years of the study.
14. Inability to provide legally effective Informed Consent Form (ICF) and/or comply with all of the required follow-up requirements
15. Subject currently participating in other investigational studies unless approved by the Sponsor in writing

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-11-13 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
PRIMARY SAFETY ENDPOINT | will be assessed up to 12-month post-procedure follow-up.
  Assess the safety of the Vivifi's Treatment through the rate & type of the procedure related complications, such as bleeding, infection or other tissue damage.
PRIMARY EFFICACY ENDPOINT | to be assessed at baseline and post-procedure 1 months, 3 months, 6 months and 12 months follow-ups.
  Assess the changes in International Prostate Symptoms Score (IPSS) from baseline to post-procedure. The score range of the questionnaire is 0 to 35. A higher score indicates worse symptomatic.

SECONDARY OUTCOMES:
SECODARY EFFICACY ENDPOINT 1 | to be assessed at baseline and post-procedure 1 months, 3 months, 6 months and 12 months follow-ups.
  Changes in International Index of Erectile Function (IIEF) questionnaire scores. The questionnaire has 15 questions. Each question is scored from 0-5. A higher score indicates improved erectile function.
SECODARY EFFICACY ENDPOINT 2 | to be assessed at baseline and post-procedure 1 months, 3 months, 6 months and 12 months follow-ups.
  Changes in size (volume) of the prostate measured by transrectal ultrasound and cystoscope in mL.
SECODARY EFFICACY ENDPOINT 3 | to be assessed at baseline and post-procedure 1 months, 3 months, 6 months and 12 months follow-ups.
  Change in peak urinary flow (Qmax) in mL/sec.
SECODARY EFFICACY ENDPOINT 4 | to be assessed at baseline and post-procedure 1 months, 3 months, 6 months and 12 months follow-ups.
  Change in post-void residual urine volume in mL.

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Starke, MD, Study Chair — Vivifi Medical (Chief Medical Officer)
Locations (1):
- Hospital Paitilla, Panama City, Provincia de Panamá, Panama